CLINICAL TRIAL: NCT06151977
Title: Impact of Lecuofiltration of Packed Red Blood Cells on Different Hematological Parameters Measured by Advia 2120
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Sayed, Doctor Yasmin, Assiut University
Other Study IDs: Leucodepleted blood parameters
Record Dates: First submitted 2023-11-16; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Leucodepletion of Packed RBC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parameters of lecuofiltration of packed Red blood cells.

DETAILED DESCRIPTION:
Impact of lecuofiltration of packed Red blood cells on different hematological parameters measured by Advia 2120

ELIGIBILITY:
Inclusion Criteria:

packed RBC ADIA2120

Exclusion Criteria:

* Whole blood

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Impact of lecuofiltration of packed Red blood cells on different hematological parameters measured by Advia 2120 | From 1/1/ 2024 to 29/12/2024
  Leucodepletion of packed RBC affects the different parameters of blood component as hemoglobin, platelets , WBCs and so on. Measurement will be done by ADIA2120 hematological analyzer by taking a sample from the packed RBC before and after leucodepletion to compare the difference in hematological parameters.

REFERENCES:
- [Background] Pandey P, Pande A, Setya D, Kumar P, Shanker A. Comparative Study for Measurement of Residual Leucocytes in Leucodepleted Red Blood Cells by Two Different Methods. Indian J Hematol Blood Transfus. 2020 Oct;36(4):740-744. doi: 10.1007/s12288-020-01325-5. Epub 2020 Aug 14. PMID 33100719